CLINICAL TRIAL: NCT00742950
Title: Study of Refractive Change Induced by 2.8-mm Corneal Incisions for Cataract Surgery
Brief Title: Refractive Change Induced by 2.8-mm Corneal Incision
Acronym: CINPHA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Jaime Tejedor / Dr, Hospital Ramón y Cajal
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CINPHACO
Record Dates: First submitted 2008-08-26; First posted 2008-08-28 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2010-05

CONDITIONS: Cataract; Refractive Surgery; Astigmatism
Keywords: Corneal incision; Cataract surgery; Phacoemulsification; Surgically induced astigmatism; Corneal Topography
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- I (Active Comparator): Nasal 2.8-mm corneal incision
  Interventions: Procedure: Nasal 2.8-mm corneal incision
- II (Active Comparator): Temporal 2.8-mm corneal incision
  Interventions: Procedure: Temporal 2.8-mm corneal incision
- III (Active Comparator): Superior 2.8-mm corneal incision
  Interventions: Procedure: Superior 2.8-mm incision

INTERVENTIONS:
Procedure: Nasal 2.8-mm corneal incision — Phacoemulsification through a nasal 2.8-mm incision
  Other Names: Phacoemulsification nasal incision
  Arms: I
Procedure: Temporal 2.8-mm corneal incision — Phacoemulsification through a 2.8-mm temporal incision
  Other Names: Phacoemulsification temporal incision
  Arms: II
Procedure: Superior 2.8-mm incision — Phacoemulsification through a superior 2.8-mm corneal incision
  Other Names: Phacoemulsification superior incision
  Arms: III

SUMMARY:
The investigators' purpose is to study the induced refractive change caused by different 2.8-mm corneal incision locations in phacoemulsification, because the investigators hypothesize that the effect may be different for nasal, temporal, and superior location, although they are considered astigmatism neutral.

Patients will be randomized to nasal or temporal incision, or assigned to superior incision, depending on preexisting astigmatism. Visual acuity, refraction, keratometry, Pentacam analysis, intraocular pressure, biomicroscopy, and funduscopy, will be carried out before and after phacoemulsification.

Outcome measures will be induced corneal refractive change (Fourier power vector analysis), ISV change, and visual acuity, at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Visual impairment for daily tasks caused by cataract
* Age older than 50 years
* Steep axis of corneal astigmatism at 90° ± 20° or 180° ± 20°
* Ability to cooperate in the protocol procedures

Exclusion Criteria:

* Age below 50
* Inability to cooperate with measurements

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Induced corneal refractive change | 6 months

SECONDARY OUTCOMES:
ISV change | 6 months
Visual acuity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Tejedor, MD, PhD, Principal Investigator — Dept Ophthalmology; José A Pérez-Rodríguez, MD, Study Chair — Dept Ophthalmology
Locations (1):
- Dept Ophthalmology, Hospital Universitario Ramón y Cajal, Madrid, Madrid, Spain

REFERENCES:
- [Background] Tejedor J, Murube J. Choosing the location of corneal incision based on preexisting astigmatism in phacoemulsification. Am J Ophthalmol. 2005 May;139(5):767-76. doi: 10.1016/j.ajo.2004.12.057. PMID 15860279
- [Derived] Tejedor J, Perez-Rodriguez JA. Astigmatic change induced by 2.8-mm corneal incisions for cataract surgery. Invest Ophthalmol Vis Sci. 2009 Mar;50(3):989-94. doi: 10.1167/iovs.08-2778. Epub 2008 Nov 14. PMID 19011013